CLINICAL TRIAL: NCT02948309
Title: Mistletoe Therapy in Primary & Recurrent Inoperable Pancreatic Cancer. A Phase III Prospective Randomized Double Blinded Multicenter Parallel Group Placebo Controlled Clinical Trial on Overall Survival and Quality of Life
Brief Title: Mistletoe Therapy in Primary and Recurrent Inoperable Pancreatic Cancer
Acronym: MISTRAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: University of Witten/Herdecke (Other); Karolinska Institutet (Other); Regional Cancer Centre Stockholm Gotland (Other); Stiftelsen Konung Gustaf V:s Jubileumsfond för cancerforskning (Unknown); Signe & Ane Gyllenbergs Stiftelse (Unknown); Ekhagastiftelsen (Other); Dagmar Ferbs Minnesfond (Unknown); Cancerforskningsfonden i Norrland (Unknown); Immunpathologisches Labor, University Tübingen (Unknown); The Sjöberg Foundation (Unknown)
Responsible Party: Principal Investigator, Kathrin Wode, MD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 131016; 2014-004552-64 (EudraCT Number)
Record Dates: First submitted 2016-09-13; First posted 2016-10-28 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer
Keywords: Primary diagnosis; Relapse
MeSH Terms: conditions — Pancreatic Neoplasms; Recurrence | interventions — viscum album peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mistletoe extract (Iscador Qu) (Experimental): Fermented aqueous extract of Viscum album ssp album (L.) (mistletoe) = Iscador Qu, subcutaneous use 3 injections/week; dose escalation from 0,01mg - 20mg
  Interventions: Drug: Mistletoe extract (Iscador Qu)
- Placebo (Placebo Comparator): isotonic saline solution, subcutaneous use 3 injections/week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mistletoe extract (Iscador Qu) — 1ml subcutaneous injection 3 times/week, dose escalation 0,01mg - 20mg
  Other Names: Fermented aqueous extract of Viscum album ssp album (L.)
  Arms: Mistletoe extract (Iscador Qu)
Drug: Placebo — 1ml subcutaneous injection 3 times/week
  Other Names: Isotonic saline solution
  Arms: Placebo

SUMMARY:
In this study a mistletoe preparation (Iscador Qu) is added to standard therapy in inoperable pancreatic cancer in order to evaluate effect on overall survival and health-related quality of life. Half of participants will take subcutaneous injections with mistletoe in addition to standard therapy (palliative chemotherapy or best supportive care); the other half will receive a placebo and standard therapy.

DETAILED DESCRIPTION:
Extracts from European mistletoe (Viscum album L.) have been used as complementary cancer therapy since the 1920s. To date over 160 clinical studies on mistletoe in cancer therapy have been conducted with varying quality; the therapy is still controversial.

Best evidence is found for increase of health-related quality of life (HRQoL) and reduction of side effects of conventional therapies (chemotherapy, radiation) in breast cancer patients. Mistletoe treatment is described as safe and well tolerated. There are some clinical studies supporting the use of mistletoe extract in the management of late stage cancer.

Statistically significant effects on overall survival (OS) and HRQoL in pancreatic cancer patients have recently been shown in a randomized open label trial in Serbia investigating the addition of mistletoe extract to best supportive care. The results are questioned because patients knew what kind of treatment they received.

Mistletoe extracts are usually administered subcutaneously. They contain a multitude of substances with immune modulatory and cytotoxic or - in animal studies - antitumorigenic, anti-metastatic and antiangiogenic effects.

This trial investigates whether there is a beneficial effect of mistletoe extracts on OS and HRQoL in pancreatic cancer patients receiving standard treatment (palliative chemotherapy or best supportive care).

Inclusion has started at 4 study centers (2 more centers are waiting for participation). And participants are randomized 1:1 to mistletoe treatment (Iscador Qu®) given in increasing dosage from 0,01mg to 20 mg or placebo injections subcutaneously 3 times /week. Stratification will be performed for received oncological treatment (palliative chemotherapy or best supportive care). At 7 visits in 9 months, participants fill in the validated EORTC QLQ-C30 (QLO=quality of life questionnaire) and PAN-26 (PAN=pancreas) quality of life questionnaires. Body weight, use of cancer-related medicines, substitution of nutrition, adverse events need of supportive care and inpatient care are measured. To be able to assess more dimensions of quality of life than possible with questionnaires, a qualitative sub-study with interviews on about 30 participants in this trial is performed in month 3. A 2nd substudy has been added november 2016 to elucidate the systemic effects of mistletoe therapy and to explore potential prognostic and predictive biomarkers (anticipated n=100).

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent

* Age ≥ 18 years
* Inoperable locally advanced or metastatic pancreatic cancer or relapse of pancreatic cancer.

  * Primary diagnosis: if histology is not clinically achievable diagnosis is to be confirmed according to local practice sufficient for diagnosis and choice of therapy (such as CA19-9 (=cancer antigen 19-9) and CT).
  * Relapse: histology (not required) or diagnosis according to local practice such as clinical signs and/or imaging and/or CA19-9.
* ECOG ( Eastern Cooperative Oncology Group) performance status 0-2 (see table in section 12.14 )
* Adequate negative pregnancy test and adequate contraception (where appropriate)

Exclusion Criteria:

Life expectancy less than 4 weeks

* Pregnancy or breastfeeding
* Neuroendocrine tumors of the pancreas (NET)
* Current use of interferon, G-CSF (granulocyte colony-stimulating factor) and thymus preparations
* Symptomatic brain edema due to brain metastases
* Known hypersensitivity to mistletoe-containing products
* Current use of mistletoe extract preparations in any form
* Chronic granulomatous disease or active autoimmune disease or autoimmune disease with immunosuppressive treatment
* Medical, psychiatric, cognitive or other conditions that may compromise the patient´s ability to understand the patient information, give informed consent, comply with the study protocol or complete the study (e.g. needle phobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2016-06; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | End of study (estimated 3 years)
  OS defined as time from randomization to death for any reason

SECONDARY OUTCOMES:
Quality of Life questionnaire EORTC QLQ-C30 | At 7 visits during study (9 months)
  Evaluation according to EORTC QLQ-C30 Scoring Manual
Quality of Life questionnaire EORTC PAN -26 | At 7 visits during study (9 months)
  Evaluation according to EORTC PAN-26 Scoring Manual
Weight in kilograms, height in meters, BMI in kg/m^2 | At 7 visits during study (9 months)
  Body weight, Body Mass Index
Corticosteroid use in milligrams betamethasone per day and indication (appetite, chemotherapy, nausea, pain, general wellbeing, other: specified) | At 7 visits during study (9 months)
  Corticosteroid use and indication
Number of visits of homecare team per week | At 7 visits during study (9 months)
  Costs for supportive care
Use of oral nutrition support per week (number used per day) | At 7 visits during study (9 months)
  Costs for supportive care
Use of symptom relieving medication in mg/day (painkillers, antiemetic and anxiolitic medication) | At 7 visits during study (9 months)
  Costs for supportive care
Chemotherapy use (number of cycles first line, second line, ..) and dose reduction in% | At 7 visits during study (9 months)
  Costs for supportive care
Number of parenteral nutrition infusions per week | At 7 visits during study (9 months)
  Costs for supportive care
Days of unplanned inpatient care | At 7 visits during study (9 months)
  Costs for inpatient care
Incidence of treatment-emergent adverse events (AE) | Through study completion (9 months)
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Annika Bergquist, Ass Prof, Study Chair — Gastrocentrum Karolinska University Hospital
Locations (1):
- Kathrin Wode, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The trial results will be submitted for publication in relevant medical journals

REFERENCES:
- [Background] Troger W, Galun D, Reif M, Schumann A, Stankovic N, Milicevic M. Quality of life of patients with advanced pancreatic cancer during treatment with mistletoe: a randomized controlled trial. Dtsch Arztebl Int. 2014 Jul 21;111(29-30):493-502, 33 p following 502. doi: 10.3238/arztebl.2014.0493. PMID 25142075
- [Background] Troger W, Galun D, Reif M, Schumann A, Stankovic N, Milicevic M. Viscum album [L.] extract therapy in patients with locally advanced or metastatic pancreatic cancer: a randomised clinical trial on overall survival. Eur J Cancer. 2013 Dec;49(18):3788-97. doi: 10.1016/j.ejca.2013.06.043. Epub 2013 Jul 24. PMID 23890767
- [Background] Horneber MA, Bueschel G, Huber R, Linde K, Rostock M. Mistletoe therapy in oncology. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD003297. doi: 10.1002/14651858.CD003297.pub2. PMID 18425885
- [Background] Kienle GS, Glockmann A, Schink M, Kiene H. Viscum album L. extracts in breast and gynaecological cancers: a systematic review of clinical and preclinical research. J Exp Clin Cancer Res. 2009 Jun 11;28(1):79. doi: 10.1186/1756-9966-28-79. PMID 19519890
- [Derived] Wode K, Kienle GS, Bjor O, Fransson P, Sharp L, Elander NO, Bernhardson BM, Johansson B, Edwinsdotter Ardnor C, Scheibling U, Hok Nordberg J, Henriksson R. Mistletoe Extract in Patients With Advanced Pancreatic Cancer: a Double-Blind, Randomized, Placebo-Controlled Tial (MISTRAL). Dtsch Arztebl Int. 2024 May 31;121(11):347-354. doi: 10.3238/arztebl.m2024.0080. PMID 38915151
- [Derived] Wode K, Hok Nordberg J, Kienle GS, Elander NO, Bernhardson BM, Sunde B, Sharp L, Henriksson R, Fransson P. Efficacy of mistletoe extract as a complement to standard treatment in advanced pancreatic cancer: study protocol for a multicentre, parallel group, double-blind, randomised, placebo-controlled clinical trial (MISTRAL). Trials. 2020 Sep 11;21(1):783. doi: 10.1186/s13063-020-04581-y. PMID 32917288